CLINICAL TRIAL: NCT05192876
Title: Analysis of Outcomes and Adverse Events of Patients Undergoing Radiation Therapy. Quality Control Using Data Base of Patient Records 2000-2025
Brief Title: Analysis of Outcomes and Adverse Events of Patients Undergoing Radiation Therapy
Status: Recruiting | Type: Observational
Sponsor: Daniel Zwahlen (Other)
Responsible Party: Sponsor-Investigator, Daniel Zwahlen, Head of Department of Radiation Oncology, Kantonsspital Winterthur KSW
Organization: Kantonsspital Winterthur KSW (Other)
Other Study IDs: BASEC-Nr. 2020-02112
Record Dates: First submitted 2021-08-04; First posted 2022-01-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Radiotherapy; Adverse Effect; Radiotherapy; Complications; Quality of Life
MeSH Terms: conditions — Radiation Injuries | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data Base of Patient Records 2000-2025: Analysis of outcomes and adverse events
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Outcomes and adverse events using radiation therapy

SUMMARY:
Analysis of outcomes and adverse events of patients undergoing radiation therapy. Quality control using data base of patient records 2000-2025

DETAILED DESCRIPTION:
What are the findings of the systematic recording and analysis of the outcomes and adverse events of radiotherapy, and how do these findings improve radiotherapy for future patients?

The goals of the systematic collection and analysis of patient-related personal data include:

* Quality assurance and showing where the quality can be improved
* Recording the outcomes and side effect profile of radiotherapy and adapting to prevent serious side effects in the future
* Presentation and publication as part of the clinical research program at the Institute for Radio-Oncology of the Winterthur Cantonal Hospital

ELIGIBILITY:
Inclusion Criteria:

* Patients who are being treated with radiotherapy at the Department of Radiation Oncology at the Winterthur Cantonal Hospital

Exclusion Criteria:

* No radiotherapy at the Department of Radiation Oncology at the Winterthur Cantonal Hospital <16 years,> 105 years

Ages: 16 Years to 105 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are being treated with radiotherapy at the Department of Radiation Oncology at the Winterthur Cantonal Hospital
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) and progression free survival (PFS) analysis after radiation therapy | 25 years
  Calculation of Overall survival (OS) and progression free survival (PFS). Time-to-event endpoints are summarized as the median and corresponding 95% confidence interval using Kaplan-Meier method
Analysis of risk factors influencing outcome after radiation therapy | 25 years
  Calculation of log-rank tests. If possible, hazard ratios are calculated via Cox regression. Competing risk analysis is conducted as supportive analysis

SECONDARY OUTCOMES:
Number of patients with acute and late adverse events after radiation therapy | 25 years
  Predefined toxicity events are described by type, grade, frequency, and percentage across all time points. Fisher's exact tests are used for comparison (base line and defined time points). Quality of life symptom and function scales are used. Two-tailed tests with a significance level of 0.05 are used for all analyses. Adjustments for multiple testing may be used. Some of the analyses are exploratory and hypothesis generating

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Zwahlen, MD, MBA, Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Windisch P, Becker I, Tang H, Schroder C, Buchali A, Aebersold DM, Zwahlen DR, Forster R, Shelan M. Converting between the International Prostate Symptom Score (IPSS) and the Expanded Prostate Cancer Index Composite (EPIC) urinary subscales: modeling and external validation. BMC Urol. 2024 Feb 3;24(1):28. doi: 10.1186/s12894-024-01421-y. PMID 38310268